CLINICAL TRIAL: NCT01237730
Title: Impact of Oropharyngeal Microorganism Colonization on the Peristomal Infection After Percutaneous Endoscopic Gastrostomy and the Effect of Tailored Antibiotics Prophylaxis
Brief Title: Tailored Antibiotics Prophylaxis for Percutaneous Endoscopic Gastrostomy
Acronym: PEG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng Kung University (Other)
Responsible Party: National cheng kung university hospital, National cheng kung univeristy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCKU-HR99
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-07

CONDITIONS: The Patients Who Receive Percutaneous Endoscopic Gastrostomy; Peristomal Wound Infection After the Operation of PEG; Prophylactic Antibiotics Before PEG
Keywords: percutaneous endoscopic gastrostomy; peristomal wound infection; prophylactic antibiotics
MeSH Terms: interventions — Cefuroxime

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cefuroxime group (Active Comparator): Use the cefuroxime as prophylactic antiobiotics, according to the clinical guideline.
  Interventions: Drug: cefuroxime
- Tailored antibiotics group (Experimental): Tailored antibiotic is selected according to the patient's oropharyngeal microorganisms.
  Interventions: Drug: Tailored antibiotic

INTERVENTIONS:
Drug: cefuroxime — Use the cefuroxime as prophylaxis.
  Arms: Cefuroxime group
Drug: Tailored antibiotic — Select the prophylactic antibiotics according to the patients oropharyngeal microorganism.
  Arms: Tailored antibiotics group

SUMMARY:
Tailored antibiotic prophylaxis according to the individual throat swab culture could reduce the peristomal infection rate

DETAILED DESCRIPTION:
Past know-how:

Antibiotic prophylaxis has been shown to be effective to reduce peristomal infection.[9-11] The penicillin-or cephalosporin-based antibiotic prophylaxis are usually used with similar efficacy.[12] EuropeanSociety of Gastrointestinal Endoscopy (ESGE) guideline recommend that a single dose of intravenous cephalosporin orpenicillin as preparation before PEG.[17] The updated practice guidelines of American Society for Gastrointestinal Endoscopy (ASGE) and British Society of Gastroenterology (BSG) also recommend cefazolin or cefuroxime as prophylactic antibiotics.[18-19]

Question:

Is the 1st or 2nd generation cephalosporin is adequate as prophylactic antibiotics for percutaneous endoscopic gastrostomy (PEG)?

Preliminary results:

1. The leading two common pathogen to cause peristomal infection of PEG are P. aeuroginosa and methecillin-resistanced S. aurous. (Figure 1) These two common pathogen can't be covered by the prophylactic antibiotics which suggested by guideline.
2. The patient with airway infection before PEG had higher peristomal infection rate, comparing with those without airway infection. Moreover, adequate antibiotics prophylaxis could significant improve the infection rate. (Table 1)

Hypothesis:

Tailored antibiotic prophylaxis according to the individual throat swab culture could reduce the peristomal infection rate.

Specific aims:

1. If individual tailored antibiotic prophylaxis according to throat swab could reduce the peristomal infection rate?
2. If the phenotype and genotype analysis were compatible between infected wound isolates and throat swab/sputum isolates?
3. If throat swab culture is better than sputum culture to predict peristomal infected microorganism?
4. Is the infection is also linked to the oropharyngeal isolates if the patients get peristomal infection more than one week after PEG?

Anticipated results:

1. Individual tailored antibiotic prophylaxis according to the throat swab culture could reduce the peristomal infection rate of PEG and short the days of hospitalization.
2. Most phenotype and genotype are compatible between peristomal isolates and throat swab/sputum isolates. It indicates that most pathogens are carried from throat into the peristomal to cause the infection. The microorganism isolated from throat swab could predict the pathogen of PEG peristomal infection.
3. The throat swab culture may be better than sputum culture to predict the peristomal infected pathogen because some unconscious patients is difficult to collect sputum.
4. Peristomal infection more than one week after PEG may be not associated to throat pathogen. It may be related to the contamination during wound care.

Significances:

This proposal result could be applied to clinical care of percutaneous endoscopic gastrostomy. The individual chose of prophylactic antibiotics could improve the peristomal infection rate. Currently, 1st or 2nd cephalosporin was usually recommended as prophylaxis before PEG. However, for the patient with ORSA culture from nasal cavity, vancomycin was suggested as prophylaxis because some studies support the benefit on infection prevention. If the results are positive, it may change the clinical guideline on antibiotics prophylaxis before PEG.

ELIGIBILITY:
Inclusion Criteria:

* The patients who receive PEG by pull method in our hospital, a tertiary transferring center, will be included

Exclusion Criteria:

* The exclusion criteria for entry are inability to place the gastrostomy for technical reasons, such as oropharyngeal deformity or esophageal stricture. The patients who receive PEG by percutaneous push method will be excluded. The patients will be also excluded if active infection and fever are identified, and the PEG is delayed until the infection is brought under control.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-07 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Peristomal wound infection | Two weeks after operation of PEG

CONTACTS AND LOCATIONS:
Overall Officials: chiao-hsiung chuang, M.D., Study Director — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan